CLINICAL TRIAL: NCT04932564
Title: Pilot Study of Leflunomide as First Line Therapy for Musculoskeletal GVHD
Brief Title: Leflunomide for Musculoskeletal GVHD After Allogeneic Stem Cell Transplant
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Issues with recruitment. Practice changes, including leflunomide use for CMV, have led to a lack of musculoskeletal GVHD cases. Only one patient enrolled in the trial will continue treatment as per standard care.
Sponsor: Tata Memorial Centre (Other)
Responsible Party: Principal Investigator, Dr Sachin Punatar, Associate Professor, Tata Memorial Centre
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 900643; CTRI/2021/04/033214 (Registry Identifier: Clinical Trials Registry- India (CTRI))
Record Dates: First submitted 2021-06-05; First posted 2021-06-21 (Actual); Last update posted 2025-09-10 (Actual); Status verified 2024-04

CONDITIONS: Musculoskeletal Disease Other; GVHD, Chronic
Keywords: Musculosceletal GVHD; Leflunomide; Allogeneic stem cell transplant
MeSH Terms: conditions — Bronchiolitis Obliterans Syndrome | interventions — Leflunomide

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Leflunomide Arm (Experimental): Leflunomide will be given at standard dose (100 mg OD x 3 days followed by 20 mg OD) in adults and weight based dose in children. This is scheduled to be continued for 1 year from the time of attaining complete response of musculoskeletal GVHD.
  Interventions: Drug: Leflunomide tablet

INTERVENTIONS:
Drug: Leflunomide tablet — Leflunomide will be given at standard dose (100 mg OD x 3 days followed by 20 mg OD) in adults and weight based dose in children.
  The dosing for children will be as follows:
  1. <20 kg - 100 mg x 1 day followed by 10 mg every alternate day
  2. 20-40 kg - 100 mg x 2 days, followed by 10 mg daily
  3. >40 kg - Usual adult dose.
  This is scheduled to be continued for 1 year from the time of attaining complete response of musculoskeletal GVHD.
  Other Names: Leflunomide

SUMMARY:
Graft versus host disease (GVHD) is a well-known complication of allogeneic transplant. In GVHD, the cells of the donor attack the patient's tissues and cause damage. It can affect any organ or system of the body. In a proportion of patients, it affects the joints and muscles. This is known as musculoskeletal GVHD. The standard treatment of musculoskeletal GVHD is steroids. However, these are usually needed for prolonged periods, and cause a large number of additional problems in transplant patients.

Leflunomide is a drug which has been used for several years in diseases like rheumatoid arthritis (RA). RA is an auto-immune disorder. The biological mechanisms underlying RA and musculoskeletal GVHD are quite similar. Hence it is likely that leflunomide may work in musculoskeletal GVHD also. The investigator have previously used leflunomide in a few patients with musculoskeletal GVHD and have found it to be extremely effective. Also, it was very safe (unlike steroids). Yet another advantage is that it is fairly cheap.

The purpose of the current study is to study the efficacy and safety of leflunomide in patients with musculoskeletal GVHD in a prospective way.

DETAILED DESCRIPTION:
The curative potential of allogeneic hematopoietic stem cell transplantation (allo-HCT) is hampered by acute and chronic graft-versus-host disease (GVHD). Although chronic GVHD (cGVHD) can affect any organ / system in the body, commonly affected are skin, oral cavity, eyes, liver, joints and fascia, and lungs. Involvement of these can occur alone or concurrently, and these lead to a significant negative impact on the patient's quality of life. Musculoskeletal involvement in chronic GVHD (mGVHD) can have varied presentations like fasciitis, myositis, arthritis, etc. The basic pathogenesis of mGvHD closely mimics autoimmune disorders like rheumatoid arthritis, systemic sclerosis, systemic lupus, etc.

The treatment goals of mGvHD include improvement or stabilisation of manifestations, limitation of long-term treatment related toxicities, improvement in functional capacity and quality of life. Corticosteroids, the standard frontline treatment, are typically administered for a median of 2 to 3years, leading to substantial morbidity. An effort to decrease corticosteroid doses has led to their use in combination with other drugs, such as cyclosporine, tacrolimus, sirolimus, mycophenolate mofetil, rituximab, etanercept, ruxolotinib, imatinib, ibrutinib, ECP (extra corporeal photopheresis), methotrexate etc, in frontline or second-line settings. All these drugs have been used with far and few responses but with significant treatment related toxicity and costs. As far as musculoskeletal GVHD is concerned, the British guidelines recommend corticosteroids as first line treatment and rituximab as second line option. However, the morbidity associated with long term steroid use warrants a quest for use of non-steroid therapies to be used in 1st line setting for chronic GVHD.

Leflunomide has been used in rheumatoid arthritis. At our centre, the investigator have previously used leflunomide for patients with musculoskeletal GVHD and found it to be effective and safe. Leflunomide is relatively cheap and potentially more effective compared to other more expensive alternatives. If proven to be effective in a larger cohort of patients, this drug could become the standard first line agent in this setting.

With this, the investigator have planned to carry out this study to assess the efficacy of leflunomide in musculoskeletal GVHD post allogeneic stem cell transplant.

ELIGIBILITY:
Inclusion Criteria:

1. Willing to give written informed consent
2. Patients diagnosed with musculoskeletal mGvHD based on 2014 NIH consensus criteria (with diagnosis confirmed by biopsy only if clinically required).
3. Willing and able to comply with all study requirements, including treatment, and periodic assessments.

Exclusion Criteria:

1. Patients with known hypersensitivity to leflunomide especially previous Steven Johnson syndrome, toxic epidermal necrolysis after leflunomide.
2. Pregnant females
3. Patients with musculoskeletal manifestations explained by other potential causes ( (drugs, trauma, etc).
4. Patients with calculated glomerular filtration rate (GFR) <30ml/min at the time of screening.

Ages: 0 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 1 (Actual)
Dates: Start 2023-09-18 (Actual); Primary Completion 2024-06-25 (Actual); Study Completion 2024-06-25 (Actual)

PRIMARY OUTCOMES:
Overall objective response rate | Through study completion, an average of 2 years
  Response will be defined as per the NIH 2014 consensus response criteria working group for mGvHD.

SECONDARY OUTCOMES:
Time to response | From date of start of leflunomide to date of first documented response, assessed up to 2 Years
  The time required to achieve complete or partial response after treatment.
Time to best response | From date of start of leflunomide to date of documented best response, assessed up to 2 Years
  Time to best response will be recorded.
Duration of response | From date of first documented response to date of first documented progression or relapse, assessed up to 2 years
  The duration of response will be calculated from the time of onset of objective response after initiation of treatment with leflunomide until the end of the follow-up, GVHD relapse, the development of new or the deterioration of pre-existing mGVHD symptoms, or the reinstitution of any additional agents to control the disease.
Relapse rate | Through study completion, an average of 2 years
  Relapse rate of mGVHD after stopping leflunomide will be recorded.

CONTACTS AND LOCATIONS:
Overall Officials: Sachin Punatar, MD, DM, Principal Investigator — Tata Memorial Centre
Locations (1):
- Tata Memorial Centre, Advanced Centre for Treatment, Research and Education in Cancer, Navi Mumbai, Maharashtra, India

IPD SHARING:
Plan to Share IPD: No